CLINICAL TRIAL: NCT03713164
Title: Exploratory Study to Determine the Bioavailability and Metabolism of Ellagic Acid From Pomegranate Juice vs. Pure Ellagic Acid
Brief Title: The Effects of Ellagic Acid From Pomegranate Juice vs. Pure Ellagic Acid on Healthy Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17-001629
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ellagic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate Juice (PJ) (Active Comparator): single dose of 8oz Pomegranate Juice (PJ)
  Interventions: Dietary Supplement: Pomegranate Juice
- Ellagic Acid (EA) (Active Comparator): 500 mg Ellagic Acid (EA) capsules
  Interventions: Dietary Supplement: Ellagic Acid

INTERVENTIONS:
Dietary Supplement: Pomegranate Juice — Volunteers will consume either one dose of pomegranate juice or pure ellagic acid, an ellagitannin naturally present in pomegranates.
  Other Names: PJ
  Arms: Pomegranate Juice (PJ)
Dietary Supplement: Ellagic Acid — Volunteers will consume either one dose of pomegranate juice or pure ellagic acid, an ellagitannin naturally present in pomegranates.
  Other Names: EA
  Arms: Ellagic Acid (EA)

SUMMARY:
The purpose of this research study is to compare the extent of polyphenol absorption in the body in normal healthy male volunteers when consuming either pomegranate juice or pure ellagic acid, an ellagitannin naturally present in pomegranates. Polyphenols are naturally occurring chemicals found in plant based food that serve to reduce inflammation and damage to cells. You will be asked to avoid foods rich in polyphenols including dark chocolate and cocoa products, dried herbs, berries, coffee, tea, flaxseeds, nuts (chestnut, hazelnut), olive and artichoke. Timed urine collections will be used to measure the metabolism of polyphenols through the presence and concentration of urolithin and ellagic acid metabolites. Additionally, it has been demonstrated in animal studies that fruits and vegetables, which are high in antioxidants and fiber, lead to improvement of gut health, inflammation and glucose tolerance. However, no information is available about the effect of ellagitanins on the gut microbiome (bacteria in the intestines).

DETAILED DESCRIPTION:
Based on the limited knowledge about the difference in bacterial metabolism of a mixture of ellagitannins, punicalin, punicalagin and EA in PJ compared to pure EA leading to intestinal formation of different urolithins (urolithin A, B and iso-urolithin A), the objective of this study is to perform a cross over acute bioavailability study of 1-day consumption of either PJ or EA. Primary endpoint will be the formation and bioavailability of EA and urolithins. Secondary endpoints will be A) effect on the fecal microbiome and B) correlation of urolithin formation to the lipid/cholesterol status of the study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years, male and any racial/ethnic group
2. Typically consume low fiber/polyphenol diet (beige diet)
3. Subjects must understand and sign the informed consent prior to participation
4. Subjects must be in generally good health
5. Subjects must be able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. Eating a high fiber/polyphenol diet or taking any medication or dietary supplements that interfere with the absorption of polyphenols.
2. History of gastrointestinal surgery, diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP > 95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
3. Screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
4. Using prebiotics, probiotics, yogurt, and/or any fiber supplements regularly
5. Allergy or sensitivity to pomegranate. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded
6. Taking antibiotics or laxatives within the past 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females have been excluded from the study to reduce the variability in the endothelial measures and Nitric Oxide determinations being performed after administration of the pomegranate or ellagic acid capsules. Estrogen is known to affect these considerably so there would be no way to control these effects among female participants in the study.
Enrollment: 19 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Compare Bioavailability of EA | 1 day
  Bioavailability of EA

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, 900 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No